CLINICAL TRIAL: NCT05723146
Title: Spatial Cognition Assessment in Virtual Reality
Acronym: CogSpa-VR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Paris Cité (Other)
Collaborators: Hopitaux de Saint-Maurice (Other); Université Paris-Saclay (Other)
Responsible Party: Principal Investigator, Alma Guilbert, Associate Professor, Université Paris Cité
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CogSpa-VR
Record Dates: First submitted 2023-01-03; First posted 2023-02-10 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Spatial Neglect
Keywords: spatial neglect; virtual reality; assessment

STUDY DESIGN:
Intervention Model Description: 60 patients with right stroke will be included in this study: a group of 30 patients with USN will be compared to a group of 30 patients without USN.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spatial cognition assessment (Experimental): A single session of spatial cognition assessment (baseline) will be proposed to participants. This assessment will be based on paper-and-pencil tasks and immersive virtual reality tasks (with an HTC Vive Pro Head-Mounted-Display). The assessment will last around 1 hour.
  Interventions: Behavioral: Spatial cognition assessment

INTERVENTIONS:
Behavioral: Spatial cognition assessment — The intervention will be composed of tasks assessing spatial cognition in a real environment (cancellation task, line bisection and baking tray task) and in a virtual environment (cancellation task, line bisection, baking tray task and localization tasks).The Catherine Bergego Scale (questionnaire) will also be used.

SUMMARY:
Unilateral spatial neglect (USN) is a highly-prevalent neuropsychological syndrome following a cerebral stroke characterized by massive impairments in daily life. The evaluation and the rehabilitation of USN encounter many limits whereas immersive virtual reality (VR) could be an efficient tool to go through these limits by imitating an environment of perception and action very close to the real one. The investigators will test a multisensory battery of evaluation based on VR for the diagnostic of USN.

ELIGIBILITY:
Inclusion Criteria:

* unilateral right stroke

Exclusion Criteria:

* epilepsy / migraine
* craniotomy
* major sensory/motor deficit
* severe cognitive impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Omissions in cancellation tasks | Baseline
  Number and localization in space
Deviation in line bisection tasks | Baseline
  Deviation of the bisection from the true center of the lines (in mm)
Number of the cubes in each side of space in the Baking Tray Tasks | Baseline
  16 cubes have to be disposed
Detections in the localization tasks | Baseline
  Number and localization in space

SECONDARY OUTCOMES:
Duration of eye fixation in each side of space during VR tasks | Baseline
  Collected thanks to the VR headset
Completion time of each task | Baseline
  (in s)
Score in the Catherine Bergego Scale (CBS) | Assessed within the same week as Baseline
  Functional assessment scored by the occupational therapists. Minimum: 0 / Maximum: 30 / Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Université Paris Cité, Paris, France

IPD SHARING:
Plan to Share IPD: No